CLINICAL TRIAL: NCT06021639
Title: Comparison of 1-day Clear Liquid Diet and Low-fiber Diet in Bowel Preparation for Colonoscopy
Brief Title: Comparison of Bowel Cleansing Regimens for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hilmi Bozkurt, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Mersin2023
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Colonoscopy Preparation
Keywords: Bowel preparation; Colonoscopy; Sennoside A+B calcium

STUDY DESIGN:
Intervention Model Description: Clear diet group (72 patients) 250 ml Sennozit A+B calcium (half dose is taken orally at 17.00 on the day before the procedure and the other half at 19.00 will be consumed. Enema 210 cc (Monobasic sodium phosphate 28.5 g. Dibasic sodium phosphate 10.5 g.) The procedure is rectal at 07.00 in the morning. will be used as Routine feeding of the patient up to the last 24 hours before the procedure. The last 24 hours will consume clear diet.
  Low fiber diet group (72 patients) 250 ml Sennozit A+B calcium (half dose is taken orally at 17.00 on the day before the procedure and the other half at 19.00 will be consumed. Enema 210 cc (Monobasic sodium phosphate 28.5 g. Dibasic sodium phosphate 10.5 g.) The procedure is rectal at 07.00 in the morning. will be used as Routine feeding of the patient up to the last 24 hours before the procedure. He/she will consume low fiber food in the last 24 hours.
Who Masked: Investigator
Masking Description: Randomization will be planned 1 to 1 according to the order of application. Randomization will be planned by the endoscopy nurse in the endoscopy unit and will not be known to the endoscopist who will perform the procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fiber diet group (Experimental): 250 ml Sennozit A+B calcium (half dose is taken orally at 17.00 on the day before the procedure and the other half at 19.00 will be consumed. Enema 210 cc (Monobasic sodium phosphate 28.5 g. Dibasic sodium phosphate 10.5 g.) The procedure is rectal at 07.00 in the morning. will be used as Routine feeding of the patient up to the last 24 hours before the procedure. He/she will consume low fiber food in the last 24 hours.
  Interventions: Dietary Supplement: The last 24 hours will consume low fiber food.
- Clear diet group (No Intervention): 250 ml Sennozit A+B calcium (half dose is taken orally at 17.00 on the day before the procedure and the other half at 19.00 will be consumed. Enema 210 cc (Monobasic sodium phosphate 28.5 g. Dibasic sodium phosphate 10.5 g.) The procedure is rectal at 07.00 in the morning. will be used as Routine feeding of the patient up to the last 24 hours before the procedure. The last 24 hours will consume clear diet.

INTERVENTIONS:
Dietary Supplement: The last 24 hours will consume low fiber food. — White bread, white rice, plain pasta or noodles, cereals not containing more than 1 gram of fiber per serving., canned or cooked skinless and seedless fruit, skinless and seedless raw fruit, pulp-free or low-fiber fruit or vegetable broth, seedless, seedless, skinless, such as canned or well-cooked carrots, string beans or peppers vegetables, tender red meat, poultry and fish, eggs, no more than two tablespoons per day, soft (creamy) peanut butter, milk, yogurt or plain cheese, salad dressings without oils or nuts, desserts without nuts.
  Arms: Low fiber diet group

SUMMARY:
Colonoscopy is a frequently used method in colon cancer screening today. Routine bowel cleansing is performed for colonoscopy. When the guidelines are examined, there are various recommendations regarding colonoscopy preparation regimens and durations. In this study, participants using the same colon cleansing drug before colonoscopy will be compared in terms of colon cleansing of the patient group who had a clear diet in the last 24 hours before the procedure and the patient group who had a low fiber diet.

DETAILED DESCRIPTION:
Studies have reported that inadequate bowel preparation reduces the detection of polyps that may have the potential to become cancerous. Unfortunately, however, many participants are unable to comply with bowel cleansing regimens due to strict dietary changes and large amounts of unpleasant laxative solutions that affect their quality of life before the procedure. In addition, participants with insufficient bowel cleansing should repeat similar preparation steps before the next examination. The European Society for Gastrointestinal Endoscopy (ESGE) recommends a polyethylene glycol (PEG) regimen for colonoscopy preparation and low-fiber food intake 24 hours prior to the procedure. In our country, PEG is not used routinely and frequently in terms of cost and lack of SGK payments. 'Sennoside A+B calcium', which is used for colonoscopy preparation in our country, shows its effect by increasing intestinal motility and causes the accumulation of water and electrolytes in the colon lumen. It has security and ease of application. In addition, the fact that it is paid by the Social Security Institution and the price is affordable makes it advantageous in the preparation of colonoscopy. Although there is not enough data for colonoscopy preparation in our country, each clinic determines the duration of the regimen in various ways. The aim of this study is to compare the patient group who used low fiber food for 24 hours before colonoscopy and who had a clear diet for 24 hours before colonoscopy in terms of adequate cleaning during endoscopy in participants who underwent bowel cleansing with 'Sennoside A+B calcium'.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Patients undergoing colonoscopy for colorectal cancer screening, or patients with nonspecific gastrointestinal symptoms

Exclusion Criteria:

* Patients with a serious medical condition such as severe heart
* Kidney or metabolic disease
* Psychiatric disease not complying with the recommended regimen
* Patients with a history of colon resection for any reason
* Patients with suspected intestinal obstruction or ileus
* Patients undergoing emergency colonoscopy
* Patients who did not accept the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Cleaning during colonoscopy | During the colonoscopy procedure
  The quality of cleaning for each segment of the colon was rated ac- cording to the Boston Bowel Preparation Scale (BBPS) as follows: Score 0 (mucosa not visible due to solid stool, or thick liquid stool cannot be cleared); Score 1 (areas of the colon segment not seen well due to staining, resid- ual stool, and/or opaque liquid); Score 2 (minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa seen well); and Score 3 (en- tire mucosa of the colon segment seen well). The left colon, transverse colon, and right colon segments were scored separately, and then these segment scores were summed for a total BBPS score ranging from 0 to 9. Categorical assessment for each possible total BBPS score: "excellent," 8-9; "good," 6-7; "fair," 5; "poor," 3-4; or "unsatisfactory," 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Hilmi Bozkurt, Principal Investigator — Mersin University
Locations (1):
- Hilmi Bozkurt, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Lorenzo-Zuniga V, Moreno-de-Vega V, Boix J. [Preparation for colonoscopy: types of scales and cleaning products]. Rev Esp Enferm Dig. 2012 Aug;104(8):426-31. doi: 10.4321/s1130-01082012000800006. Spanish. PMID 23039803
- [Background] Ozer Etik D, Suna N, Gunduz C, Bostan A, Ozdemir A, Gurel BY, Yenisekerci E, Boyacioglu AS. Can a 1-day clear liquid diet with a split -dose polyethylene glycol overcome conventional practice patterns during the preparation for screening colonoscopy? Turk J Gastroenterol. 2019 Sep;30(9):817-825. doi: 10.5152/tjg.2019.19071. PMID 31258137
- [Background] Labianca R, Merelli B. Screening and diagnosis for colorectal cancer: present and future. Tumori. 2010 Nov-Dec;96(6):889-901. PMID 21388049
- [Background] Haseman JH, Lemmel GT, Rahmani EY, Rex DK. Failure of colonoscopy to detect colorectal cancer: evaluation of 47 cases in 20 hospitals. Gastrointest Endosc. 1997 Jun;45(6):451-5. doi: 10.1016/s0016-5107(97)70172-x. PMID 9199899
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Faiss S. The missed colorectal cancer problem. Dig Dis. 2011;29 Suppl 1:60-3. doi: 10.1159/000331119. Epub 2011 Nov 15. PMID 22104756